CLINICAL TRIAL: NCT06546943
Title: Glucose Monitoring in Youth With Cystic Fibrosis During Pulmonary Exacerbations (GeM-PEx)
Brief Title: Glucose Monitoring in Youth With Cystic Fibrosis During Pulmonary Exacerbations
Acronym: GeM-PEx
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 21-3666
Record Dates: First submitted 2023-11-08; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cystic Fibrosis Pulmonary Exacerbation
Keywords: cystic fibrosis related diabetes; continuous glucose monitoring; cystic fibrosis pulmonary exacerbation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — optional blood sampling to run inflammatory markers at end of study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study is to investigate the prevalence of dysglycemia with continuous glucose monitoring (CGM) obtained during pulmonary exacerbations, both outpatient and inpatient, in youth with cystic fibrosis (CF).

DETAILED DESCRIPTION:
This research is using continuous glucose monitoring (CGM) to study changes in blood sugar levels that may occur in youth with cystic fibrosis (CF) and cystic fibrosis related diabetes (CFRD) who experience a pulmonary exacerbation (PEx), whether admitted to the hospital or seen in clinic. We hypothesize that 1) youth experiencing a PEx will have greater blood sugar changes during the PEx than at least 6 weeks after the PEx , 2) that the changes in blood sugars will be greater during the PEx when compared to CGM data gathered at a baseline visit prior to the PEx (when available), 3) and that blood sugar changes during the PEx will compare with changes in short-term clinical outcomes collected using questionnaires about breathing problems, and that this data will be predictive of the need for additional antibiotics. This study aims to compare CGM measures of change during a PEx with those measured after recovery; to compare CGM measures of change during the PEx to those taken at baseline; and to examine the relationships between these changes and the changes in clinical findings including the need for additional antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* 6- 25 years old
* Confirmed diagnosis of cystic fibrosis (based on sweat chloride and/or two known disease causing CF mutations)
* access to a smart phone and/or internet connection and the ability to complete remote telehealth visits

Exclusion Criteria:

* known type 1 or type 2 diabetes, monogenic diabetes
* critical illness requiring admission to the ICU
* pregnancy

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals with CF ages 6 y- 25 years will be eligible to enroll. Participants will be enrolled at baseline health during a routine CF clinic visit or upon diagnosis of a pulmonary exacerbation (PEx). A PEx will be defined by treatment with either oral or IV antibiotics for an increase in respiratory symptoms as defined by a pediatric pulmonologist at our CF Center. Oral antibiotics are typically prescribed for two weeks based on clinical care guidelines developed at our center which standardize antibiotic selection based on prior respiratory culture results.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
CGM standard deviation | 14 days
  Measures of glycemic variability from CGM during the exacerbation (CGM-PEx) compared measure derived from recovery period (CGM-post)
CGM coefficient of variation | 14 days
  CGM measure of glycemic variability during the exacerbation (CGM-PEx) with recovery measure (CGM-post)
MAGE (mean amplitude of glycemic excursions) | 14 days
  CGM measures of glycemic variability (MAGE) during the exacerbation (CGM-PEx) with recovery measures (CGM-post)

SECONDARY OUTCOMES:
Forced expiratory volume at one second (FEV1) at each visit | up to 2 years
  Collected clinically at baseline during routine visits, and at the start of a pulmonary exacerbation (PEx) for those admitted inpatient and in clinic, and at next in person routine clinic visit; b)by home spirometer during routine clinic visits, and in the hone setting (if not in person) once for the baseline visit, and at the onset of exacerbation and twice/week for 14 days, and once upon recovery (at least 6 weeks after PEx)
Need for additional antibiotics within 28 days following initial treatment | up to 2 years
  If initial Rx for antiobiotics proves unsuccessful and participant requires additional treatment
Chronic Respiratory Infection Symptom Score questionnaire | up to 2 years
  Questionnaire tracking exacerbation symptoms
sputum culture as available from clinical data | up to 2 years
  Will be collected when available from clinical data
markers of inflammation when available | up to 2 years
  hsCRP (highly sensitive C-Reactive Protein) and cytokines (eg; Interleukin-6 [IL 6] & Interleukin-8 [IL8]) at visits
Cystic Fibrosis Questionnaire Revised (CFQR) questionnaire | up to 2 years
  quality of life questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, University of Colorado Denver, Aurora, Colorado, United States